CLINICAL TRIAL: NCT05818150
Title: Multicenter, PrOspective, Randomized, Controlled Trial Comparing GenIcular Artery EmbOlization Using Embosphere Microspheres to Corticosteroid iNjections for the Treatment of Symptomatic Knee Osteoarthritis: MOTION Study
Brief Title: GAE Using Embosphere Microspheres vs Corticosteroid Injections for Treatment of Symptomatic Knee OA (MOTION)
Acronym: MOTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAE-P3-22-01
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis
Keywords: genicular artery embolization; GAE; knee embolization; knee OA
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones; Triamcinolone; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomized 1:1 to either geniculate artery embolization or corticosteroid injection for treatment of symptomatic knee osteoarthritis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Genicular artery embolization with Embosphere Microspheres (Experimental): Device: Embosphere Microspheres
  Embolic Agent: Embosphere Microspheres
  Interventions: Device: Embosphere Microspheres
- Corticosteroid Injection of the knee (Active Comparator): Drug: Corticosteroid injection
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Device: Embosphere Microspheres — Embolic Agent: Embosphere Microspheres
  Other Names: Genicular artery embolization
  Arms: Genicular artery embolization with Embosphere Microspheres
Drug: Corticosteroid injection — Corticosteroid injection
  Other Names: Triamcinolone or methylprednisolone
  Arms: Corticosteroid Injection of the knee

SUMMARY:
This multicenter, prospective, interventional trial is designed to assess the outcome of subjects with symptomatic knee osteoarthritis (OA) that are randomized to treatment with either genicular artery embolization (GAE) using Embosphere Microspheres or steroid injection over a period of 24 months.

DETAILED DESCRIPTION:
This study is an IDE study. It is an RCT comparing GAE to steroid injection in the knee to treat knee osteoarthritis.

ELIGIBILITY:
Key Inclusion Criteria:

Provides written informed consent

Age ≥21 years

Mild to severe knee pain, defined as a WOMAC Pain score of ≥8 out of 20 (in the target knee)

Pain refractory to conservative therapies for at least 90 days prior to enrollment/randomization.

Kellgren-Lawrence grade 1, 2, 3 or 4

Key Exclusion Criteria:

Planned major surgical or endovascular procedures ≤ 30 days after the index procedure.

Advanced atherosclerosis

Known history of rheumatoid or infectious arthritis.

Prior knee replacement surgery of the target knee.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 6 months
  Clinical Success defined as ≥50% improvement in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale from baseline to 6 months without the need for additional intervention.
Primary Safety Endpoint | 6 months
  Freedom from treatment-related safety events through 6 months (180 days) following the index procedure.

SECONDARY OUTCOMES:
Subjects achieving Clinical Success | 3, 12, and 24 months
  Number of subjects achieving Clinical Success
Numerical rating scale (NRS) | baseline, 3, 6, 12 and 24 months
  Pain score assessed using numerical rating scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Bagla, MD, Principal Investigator — Prostate Centers, USA; Craig J McAsey, MD, Principal Investigator — Anderson Orthopedic Clinic
Locations (27):
- United States (19):
  - Memorial Care Long Beach Medical Center, Long Beach, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Biotech Clinical Research/ Georgia Vascular Institute, College Park, Georgia
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Saint Louis University, St Louis, Missouri
  - Atlantic Medical Imaging, Galloway, New Jersey
  - Rutgers Health, Newark, New Jersey
  - Northwell Health, Manhasset, New York
  - Weill Cornell Medicine, New York, New York
  - Atlas Interventional, Williamsville, New York
  - Prostate Centers USA, Raleigh, North Carolina
  - Sunrise Vascular Center, Sanford, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Cardiovascular Health Clinic, Oklahoma City, Oklahoma
  - Prostate Centers USA, Falls Church, Virginia
  - Prostate Centers USA, Leesburg, Virginia
- Liverpool Hospital, Liverpool, Australia
- Brazil (2):
  - Hospital de Clínicas de Passo Fundo, Passo Fundo
  - University of Sao Paulo, São Paulo
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - CHUM - Centre hospitalier de l'Université de Montréal, Montreal
- North Shore Hospital/ Te Whatu Ora - Waitemata, Takapuna, New Zealand
- United Kingdom (2):
  - University Hospitals Dorset, Bournemouth
  - Grange University Hospital, Cwmbran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bent C, McAsey CJ, Bagla S. Multicenter, PrOspective, Randomized, Controlled Trial Comparing GenIcular Artery EmbOlization Using Embosphere Microspheres to Corticosteroid iNjections for the Treatment of Symptomatic Knee Osteoarthritis: MOTION Study Protocol Summary. Cardiovasc Intervent Radiol. 2025 Apr;48(4):551-558. doi: 10.1007/s00270-025-03994-z. Epub 2025 Mar 6. PMID 40050421